CLINICAL TRIAL: NCT04922944
Title: Post Vaccination Antibody Assays and Reactions in Hospital Employees and Medical Staff: an Analysis of Antibody Response Over Time
Brief Title: Post COVID-19 Vaccination Analysis in Healthcare Worker Recipients
Status: Completed | Type: Observational
Sponsor: Huntington Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00050032
Record Dates: First submitted 2021-03-30; First posted 2021-06-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Covid19; Vaccine Reaction
Keywords: SARS-CoV-2; vaccination; antibody formation
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: COVID-19 vaccine — Two-dose COVID-19 vaccine
  Other Names: Pfizer-BioNTech COVID-19 vaccine; Moderna COVID-19 vaccine

SUMMARY:
This research study is studying how healthcare worker recipients react after receiving vaccinations for COVID-19. The objective of the study is to evaluate the immune response to COVID-19 vaccination. The immunity will be evaluated over time by measuring serum semi-quantitative SARS-Co-V2 IgG from blood specimens and analyzing vaccine reaction data. SARS-CoV-2 is the name for the virus responsible for COVID-19 infections. IgG, immunoglobulin G, is an antibody found in the blood that protects against bacterial and viral infections. Study subjects will also be asked to report physical reactions they may have experienced related to vaccinations.

DETAILED DESCRIPTION:
As some of the first recipients of SARS-CoV-2 vaccines under emergency authorization use, healthcare workers represent a diverse subpopulation, that are now moving through the immune response to the Pfizer and Moderna mRNA vaccines. As individual responses may vary, this provides an opportunity to evaluate levels of IgG response in relation to age, gender, comorbidities and other factors that may influence immunity. We recognize that, though this is only part of the immune response that may be protective for severe COVID-19 disease, it is a first step in understanding the level and durability of post vaccination SARS-CoV-2 antibodies.

This small, pilot study will evaluate the immune response over time by measuring serum semi-quantitative SARS-CoV-2 IgG from healthcare vaccinees at various timepoints. A high-level review of reactions related to the vaccinations will be performed with the same population of healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for study
* Current employee or active member of the medical staff of Huntington Hospital, Pasadena, CA, (must have valid hospital identification)
* Must have completed vaccination regimen (two doses if required) no more than 8 weeks ± 5 days before enrollment
* Must have completed, valid vaccination card, if vaccinations received at a center other than Huntington Hospital
* Able to read English, sign consent form and complete on-line surveys

Exclusion Criteria:

* Huntington Hospital employees on leave of absence
* Anyone not able/willing to provide blood specimens and respond to surveys for the 52-week study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Current employee or active member of the medical staff of Huntington Hospital, Pasadena, CA who has completed the vaccination regimen
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in SARS-CoV-2 IgG Titer Over Time | 8 weeks (± 5 days) post-vaccination regimen completion; 24 weeks (± 5 days) post-vaccination regimen completion; and 52 weeks (± 5 days) post-vaccination regimen completion
  Semi-quantitative SARS-CoV-2 IgG titer

SECONDARY OUTCOMES:
Occurrence of post-vaccine reactions | Within 3 days after vaccine injections
  Subjective reporting of occurrence of post-vaccination reactions including anaphylactic reactions (such as difficulty breathing, swelling of face and throat, fast heartbeat, bad rash all over body, and dizziness and weakness); injection site pain; injection site swelling/hardness; injection site redness; tiredness; headache; muscle pain; chills; join pain; fever; nausea; feeling unwell; and/or swollen lymph nodes
Severity of post-vaccine reactions | Within 3 days after vaccine injections
  Subjective reporting of severity of post-vaccine reactions (none, mild, moderate, or severe)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Shriner, MD, Principal Investigator — Huntington Hospital
Locations (1):
- Huntington Hospital, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No